CLINICAL TRIAL: NCT06204445
Title: Exploratory Study of the Interindividual Variation in Response to Consumption of a Polyphenol-rich Green Coffee and Factor Influencing the Response
Brief Title: Interindividual Variation in Response to Green Coffee
Acronym: GREENCOF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PID2020-114102RB-I00
Record Dates: First submitted 2023-12-30; First posted 2024-01-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
Keywords: Inter-individual variability; (Poly)phenols; Green coffee; Obesity; Genotype; Microbiota; Bioavailability and metabolism; Lifestyle; Cardiometabolic and inflammatory biomarkers
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: After a run-in period, participants are randomly allocated to one of each arm. Each intervention last 12 weeks, separated by a 4-week wash-out.
Who Masked: Participant, Outcomes Assessor
Masking Description: Coffee is provided as ground coffee in unmarked 1 kg packets labeled A or B for blinding, with instructions on how to prepare the coffee brew. The polyphenol-rich coffee is slightly roasted to emulate flavor, color and aroma for blinding.
  Assessor will only be presented results marked as intervention A and B. Only the PIs will know the order in which both coffees were consumed by volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Green (slightly roasted) coffee (Experimental): Slightly roasted ground Arabica coffee rich in phenolic compounds (hydroxycinnamic acids). Participants will consume 3 cups of freshly brewed coffee daily (breakfast, mid-morning, early afternoon). Black coffee, no milk.
  Interventions: Dietary Supplement: Green coffee
- Roasted coffee (Active Comparator): Traditional roasted ground coffee (Arabica). Participants will consume 3 cups of freshly brewed coffee daily (breakfast, mid-morning, early afternoon). Black coffee, no milk.
  Interventions: Dietary Supplement: Roasted coffee

INTERVENTIONS:
Dietary Supplement: Green coffee — Each cup of coffee provides approximately 400 mg of hydroxycinnamic acids.
  Arms: Green (slightly roasted) coffee
Dietary Supplement: Roasted coffee — Each cup of coffee provides approximately 150 mg of hydroxycinnamic acids.
  Arms: Roasted coffee

SUMMARY:
The study is a multifaceted approach to investigate the effects of regular consumption of green coffee rich in polyphenols (hydroxycinnamic acids) on weight, body composition, cardiometabolic and inflammatory biomarkers in a sample population of overweight and obese people aimed at identifying a population of responders to green coffee experimenting the highest benefit from this product, and to contribute to the understanding of the influence of some of the main factors on the response to green coffee and their association with the differences between individuals (high-responders vs. low-responders).

DETAILED DESCRIPTION:
A randomized, cross-over, blind clinical trial will be carried out to evaluate the health effects of a polyphenol-rich green (slightly roasted) coffee in comparison with traditional roasted coffee to identify high- and low-responders.

Participants will consume the green and roasted coffee in a randomized order during 12 weeks, separated by a 4-week wash-out (and a previous 2-week run-in). Fasting blood samples will be collected in each of the 6 visits to the research centre. Blood pressure and body composition and anthropometric variables will be measured. In addition, urine and fecal samples will be obtained at the beginning and end of each intervention stage to analyze the bioavailability and metabolism of phenolic compounds, and the intestinal microbiota, respectively. Physical activity and energy expenditure will be measured in each of the interventions.

Besides a thorough cardiometabolic and inflammatory characterization of the volunteers, the frequency of specific genotypes (related with obesity, energy metabolism, inflammation and coffee intake) will be analyzed, as well as lifestyle and dietary habits of the participants, including aspects such as chrono-nutrition, sleep quality and wellbeing perception with the aim to contribute to clarify the determinants of inter-individual variability in the health effects of coffee bioactive phenolic compounds.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25-35 kg/m2

Exclusion Criteria:

* Smoking
* Vegetarian/Vegan
* Pregnant/lactating women
* On prescription drugs other than for thyroid/hypertension/dyslipemia, or changes in dosage in the last 3 months.
* Consumption of vitamins or dietary supplements
* On weight-reduction dietary regime or physical training to reduce body weight
* Having taken antibiotics 3 months before starting the intervention
* Intestinal, hepatic or renal diseases, coffee intolerance

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Body weight | 12-week
  Change in body weight (estimated 2.5 kg) at the end of the intervention
Body fat percentage | 12 weeks
  Change in body fat percentage (total and visceral) at the end of the intervention

SECONDARY OUTCOMES:
Blood lipids | 12 weeks
  Change in serum levels of total cholesterol or LDL-cholesterol, HDL-cholesterol or triglycerides at the end of the intervention
Blood glucose | 12 weeks
  Change in fasting blood glucose levels at the end of the intervention
Insulin levels | 12 weeks
  Change in fasting blood insulin levels at the end of the intervention
Insulin resistance | 12 weeks
  Change in homeostasis model assessment (HOMA) of insulin resistance (HOMA-IR) index at the end of the intervention
Insulin sensitivity | 12 weeks
  Change in quantitative insulin sensitivity check index (QUICKI) at the end of the intervention.
Glycated hemoglobin | 12 weeks
  Change in blood levels of glycated hemoglobin (HbA1c) at the end of the intervention
Inflammatory cytokines | 12 weeks
  Change in the levels of the pro-inflammatory cytokines tumor necrosis factor-alpha (TNFa), interleukin (IL)-1beta, IL-2, IL-6, or anti-inflammatory IL-10 at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bravo, Prof, Principal Investigator — Instituto de Ciencia y Tecnología de Alimentos y Nutrición
Locations (1):
- Instituto de Ciencia y Tecnología de Alimentos y Nutrición, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Interested researchers may contact the principal investigator.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After completion of the study and publication of results
Access Criteria: Justified request to the principal investigator